CLINICAL TRIAL: NCT00866034
Title: Prospective, Multicenter,Randomized Controlled Trial Towards Identifying the Optimal GnRH Antagonist Treatment Protocol
Brief Title: Cetrotide Treatment Optimization
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to limited rate of patient inclusion
Sponsor: Bart CJM Fauser (Other)
Responsible Party: Sponsor-Investigator, Bart CJM Fauser, Professor of Reproductive Medicine and Gynecology, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CETRO Trial; CCMO: NL23973.041.08; METC: 08-262/G-K
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: In Vitro Fertilization; Intracytoplasmic Sperm Injection
Keywords: Cetrotide; IVF; ICSI; Treatment protocol
MeSH Terms: interventions — cetrorelix; Ovulation Induction; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD2 (Experimental): Early fixed start of a daily dose of 0.25mg Cetrotide on cycle day 2, together with the initiation of daily treatment with exogenous gonadotropins.
  Interventions: Drug: Cetrotide (Ovarian stimulation)
- CD6 (Experimental): Late fixed start of a daily dose of 0.25mg Cetrotide on cycle day 6. As in the other arm of the study, exogenous gonadotropins will commence on cycle day 2.
  Interventions: Drug: Cetrotide (Ovarian stimulation)

INTERVENTIONS:
Drug: Cetrotide (Ovarian stimulation) — Fixed start of a daily dose of 0.25mg Cetrotide on cycle day 2
  Other Names: Gonal-F; Cetrorelix
  Arms: CD2
Drug: Cetrotide (Ovarian stimulation) — Late fixed start of a daily dose of 0.25mg Cetrotide on cycle day 6.
  Other Names: Gonal-F; Cetrorelix
  Arms: CD6

SUMMARY:
Rationale:

In daily practice fertility treatment is increasingly patient focused and innovative medication and standardized treatment guidelines are being developed to improve patient convenience.

GnRH antagonist cotreatment to prevent premature luteinization during ovarian stimulation for IVF and ICSI greatly reduces the burden of treatment, partly by reducing the number of injections by around 21 compared with the optimal GnRH agonist 'long' protocol. However, the optimal GnRH antagonist protocol is still not known. There are a number of reasons to suggest that both the simplicity of treatment and clinical outcomes could be further improved by commencing GnRH antagonist treatment on the same day on which ovarian stimulation is started. These include more synchronized follicle development and reduced rates of premature luteinization. This study will investigate whether a novel early fixed start protocol improves outcomes in comparison to the widely employed late fixed start protocol.

Objective:

To demonstrate whether an early fixed start antagonist protocol improves the live birth rate compared with a late fixed start antagonist protocol by 5%.

Study design:

Prospective, multicenter, investigator sponsored, randomized controlled trial

Study population:

* Normo-ovulatory women < 39 years with an indication for IVF or ICSI
* No more than 2 previous unsuccessful IVF/ICSI cycles
* BMI ≤ 32 kg/m2

Intervention:

Two different GnRH antagonist treatment protocols used in daily practice will be compared. Patients will be randomized to receive one of the following two treatments:

* Early fixed start: start GnRH antagonist treatment with Cetrotide 0.25 mg on the same day as FSH, cycle day 2.
* Late fixed start: FSH will be administered from cycle day 2. GnRH antagonist treatment with Cetrotide 0.25 mg will commence on cycle day 6.

Main study parameters/endpoints:

The primary endpoint is the live birth rate per started cycle. A secondary endpoint is the number of embryos available for transfer.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

In addition to recording clinical outcomes, endocrine studies will be carried out at the UMC Utrecht in a sample of 200 participants who will be subjected to blood sampling at three points during the treatment cycle: prior to commencing treatment on cycle day 2, cycle day 6 and the day of hCG administration.The aim of this substudy was therefore to prospectively compare the effect of a cycle day 2 versus cycle day 6 fixed start GnRH antagonist protocol on LH, estradiol and progesterone levels in the mid and late follicular phase. In order to investigate whether the early fixed protocol exerts a significant extra burden on patients compared to the late start protocol, another group of 200 participants at the UMCU will be requested to complete the HADS questionnaire (Hospital Anxiety and Depression Scale).

ELIGIBILITY:
Inclusion Criteria:

* Normo-ovulatory women < 39 years with an indication for IVF or ICSI

Exclusion Criteria:

* More than 2 previous unsuccessful IVF/ICSI cycles
* BMI > 32 kg/m2

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 617 (Actual)
Dates: Start 2009-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick S Macklon, Prof, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Hamdine O, Macklon NS, Eijkemans MJ, Laven JS, Cohlen BJ, Verhoeff A, van Dop PA, Bernardus RE, Lambalk CB, Oosterhuis GJ, Holleboom CA, van den Dool-Maasland GC, Verburg HJ, van der Heijden PF, Blankhart A, Fauser BC, Broekmans FJ; CETRO trial study group. Elevated early follicular progesterone levels and in vitro fertilization outcomes: a prospective intervention study and meta-analysis. Fertil Steril. 2014 Aug;102(2):448-454.e1. doi: 10.1016/j.fertnstert.2014.05.002. Epub 2014 Jun 11. PMID 24929258
- [Derived] Hamdine O, Macklon NS, Eijkemans MJ, Laven JS, Cohlen BJ, Verhoeff A, van Dop PA, Bernardus RE, Lambalk CB, Oosterhuis GJ, Holleboom CA, van den Dool-Maasland GC, Verburg HJ, van der Heijden PF, Blankhart A, Fauser BC, Broekmans FJ; CETRO trial study group. Comparison of early versus late initiation of GnRH antagonist co-treatment for controlled ovarian stimulation in IVF: a randomized controlled trial. Hum Reprod. 2013 Dec;28(12):3227-35. doi: 10.1093/humrep/det374. Epub 2013 Oct 15. PMID 24129613
- [Derived] Hamdine O, Broekmans FJ, Eijkemans MJ, Lambalk CB, Fauser BC, Laven JS, Macklon NS; CETRO trial study group. Early initiation of gonadotropin-releasing hormone antagonist treatment results in a more stable endocrine milieu during the mid- and late-follicular phases: a randomized controlled trial comparing gonadotropin-releasing hormone antagonist initiation on cycle day 2 or 6. Fertil Steril. 2013 Sep;100(3):867-74. doi: 10.1016/j.fertnstert.2013.05.031. Epub 2013 Jun 27. PMID 23809501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 2009 - July 2011 Six hundred and seventeen women undergoing IVF or ICSI were recruited from the IVF outpatient clinics of 13 fertility centres.
Pre-assignment Details: None were excluded before assignment.
Groups:
- Early Start CD2: Early fixed start of a daily dose of 0.25mg Cetrotide on cycle day 2, together with the initiation of daily treatment with exogenous gonadotropins.
- Late Start CD6: Late fixed start of a daily dose of 0.25mg Cetrotide on cycle day 6. As in the other arm of the study, exogenous gonadotropins will commence on cycle day 2.
Period: Overall Study
Arm/Group | Early Start CD2 | Late Start CD6
Started | 308 | 309
Completed | 292 | 301
Not Completed | 16 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Start CD2 | Late Start CD6 | Total
Number analyzed (Participants) | 308 | 309 | 617
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 308 | 309 | 617
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (3.9) | 32.2 (4.2) | 32.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308 | 309 | 617
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 308 | 309 | 617

OUTCOME MEASURES:

1. Primary Outcome: Live Birth Rate Per Started Cycle and Live Birth From Cryopreserved Embryos Originating From, and Occurring Within 6 Months of the Initial Treatment Cycle Will be Included in the Total Live Birth Rate Per Started Cycle.
Time Frame: 2 years
Measure: Number; unit: Cumulative live birth rate (%)
Arm/Group | Early Start CD2 | Late Start CD6
Number analyzed (Participants) | 308 | 309
Cumulative live birth rate (%) | 26.7 | 29.9

2. Secondary Outcome: Cumulative Ongoing Pregnancy Rate
Time Frame: 2 years
Measure: Number; unit: cumulative ongoing pregnancy rate (%)
Arm/Group | Early Start CD2 | Late Start CD6
Number analyzed (Participants) | 308 | 309
cumulative ongoing pregnancy rate (%) | 27.6 | 31.4

3. Other Pre Specified Outcome: Endocrine Profile in the Early, Mid and Late Follicular Phase.
Description: 1. difference in endocrine profile between the 2 arms during the mid and late follicular phase
  2. influence of early elevated follicular phase progesterone levels on clinical outcome
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Early Start CD2 | Late Start CD6
Serious Adverse Events (participants affected / at risk) | 4/308 | 8/309
Other Adverse Events (participants affected / at risk) | 20/308 | 18/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Start CD2 (N=308) | Late Start CD6 (N=309)
OHSS (Reproductive system and breast disorders) | 4 (4) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Start CD2 (N=308) | Late Start CD6 (N=309)
cancellation due to hyperresponse (Reproductive system and breast disorders) | 7 (7) | 3 (3)
cancellation due to hyporesponse (Reproductive system and breast disorders) | 13 (13) | 15 (15)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely because no significant difference was observed in clinical outcome after 617 inclusions. A much larger population would be needed to detect a small significant difference in favour of either study arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No